Study: # 7280 entitled Treatment of Cannabis Use Disorder among adults with co-morbid Attention-Deficit/Hyperactivity Disorder

PI: Frances R. Levin

NCT# NCT02803229

Study Protocol Date: June 07, 2016

#### **New York State Psychiatric Institute**

### **Institutional Review Board**

June 7, 2016

| To: | Dr. | Frances | R. | Levin |
|-----|-----|---------|----|-------|

**From**: Dr. Edward Nunes, Co-Chairman

Dr. Laurence Greenhill, Co-Chairman

**Subject:** APPROVAL NOTICE

Your protocol #7280 entitled: TREATMENT OF CANNABIS USE DISORDER AMONG ADULTS WITH COMORBID ATTENTION-DEFICIT/HYPERACTIVITY DISORDER (version date 06-07-16) and consent form have been approved by the New York State Psychiatric Institute - Columbia University Department of Psychiatry Institutional Review Board from June 7, 2016 to April 3, 2017 (Reviewed by the Full Board on 04-04-16).

| Consent requirements: |
|---|
| $\square$ Not applicable |
| ☐ 45CFR46.116(d) waiver or alteration of consent for the telephone interview |
| X Signature by the person(s) obtaining consent is required to document the consent process. |
| ☐ Documentation of an independent assessment of the participant's capacity to consent is also required. |
| Approved for recruitment of subjects who lack capacity to consent: ${f X}$ No $\Box$ Yes |
| Field Monitoring Requirements: X Routine □ Special: |

- ✓ Only copies of consent documents that are currently approved by the IRB may be used to obtain consent for participation in this study.
- ✓ A progress report and application for continuing review is required 2 months prior to the expiration date of IRB approval.
- ✓ Changes to this research may not be initiated without the review and approval of the IRB except when necessary to eliminate immediate hazards to participants.
- ✓ All serious and/or unanticipated problems or events involving risks to subjects or others must be reported immediately to the IRB. Please refer to the PI-IRB website at <a href="http://irb.nyspi.org">http://irb.nyspi.org</a> for Adverse Event Reporting Procedures and additional reporting requirements.

Enc: CF, HIPAA form

CC: RFMH Business Office (U54DA037842-01)

**CU Grants & Contracts** 

**CUMC-IRB** 

EN/LG/Scr

### NEW YORK STATE PSYCHIATRIC INSTITUTE INSTITUTIONAL REVIEW BOARD

Levin, Frances

Protocol Title: Version Date: Treatment of Cannabis Use Disorder 06/07/2016

among Adults with Comorbid Attention-

**Deficit/Hyperactivity Disorder** 

Protocol Number:

7280

Clinic:

**Substance Treatment And Research** First Approval:

06/07/2016 Services (STARS)

**Expiration Date:** 04/03/2017

Principal Investigator: Co-Investigator(s): Frances Levin, MD John Mariani, MD

Email: frl2@columbia.edu

**Telephone:** 646-774-6137

Research Chief: Frances Levin, MD

#### **Cover Sheet**

Choose from the following that is applicable to your study I am submitting a new protocol

#### **Division & Personnel**

#### **Division**

What Division/Department does the PI belong to? Substance Use

Within the division/department, what Center or group are you affiliated with, if any?

**STARS** 

#### **Unaffiliated Personnel**

List investigators, if any, who will be participating in this protocol but are not affiliated with New York State Psychiatric Institute or Columbia University. Provide: Full Name, Degrees and Affiliation. This project is a single-site trial.

#### **Procedures**

### To create the protocol summary form, first indicate if this research will include any of the following procedures

- ✓ Psychiatric Assessment
- ✓ Collection of Biological Specimens
- ✓ Medication Trial
- ✓ Use of Placebo or Sham Treatment
- ✓ Medication-Free Period or Treatment Washout
- ✓ Off-label Use of Drug or Device
- ✓ Internet-based Data Collection or Transmission

### **Population**

#### Indicate which of the following populations will be included in this research

- Medically and Psychiatrically Healthy Subjects
- ✓ Adults
- ✓ Adults over 50
- ✓ Substance Users

### **Research Support/Funding**

Will an existing internal account be used to support the project?

Yes

Describe internal account

U54DA037842-01 Shared Pharmacotherapeutic Strategies for Cannabinoid & Opioid Use Disorders

Is the project externally funded or is external funding planned?

Yes

Select the number of external sources of funding that will be applicable to this study

#### Funding Source #1

Is the PI of the grant/contract the same as the PI of the IRB protocol?

Yes

Select one of the following

The grant/contract is currently funded

Source of Funding

Federal

Institute/Agency

NIDA

Grant Name

Shared Pharmacotherapeutic Strategies for Cannabinoid & Opioid Use Disorders

Grant Number

U54DA037842-01

Select one of the following

Single Site

**Business Office** 

**RFMH** 

Does the grant/contract involve a subcontract?

Yes

Subcontracted?

To

Name institution(s)

Columbia University

### **Study Location**

Indicate if the research is/will be conducted at any of the following

✓ NYSPI

✓ Other Columbia University Medical Center Facilities

This protocol describes research conducted by the PI at other facilities/locations

Yes

✓ Hospital, clinics and other healthcare facilities

#### Hospitals, clinics and other healthcare facilities

Select from the list

or type in location(s)...

STARS at Columbia University, 3 Columbus Circle, 14th floor, Suite 1403

### Lay Summary of Proposed Research

Lay Summary of Proposed Research

The proposed protocol is a double-blind, placebo-controlled outpatient study of the safety and benefit of Extended-release mixed amphetamine salt (Adderall-XR, MAS-XR) in the treatment of individuals with CUD and ADHD. We plan to randomize 40 patients in a 12-week trial. The primary objective of the study is to determine the efficacy of MAS-XR in promoting cannabis abstinence among individuals with CUD and in promoting a decrease of ADHD symptoms.

### Background, Significance and Rationale

Background, Significance and Rationale

ADHD is common in substance use disorder patients in general and cannabis use disorder (CUD) in

Protocol Summary Form 7280 Levin, Frances

particular, occurring at rates substantially greater than in the general population. A meta-analysis found that approximately 23% of substance abusers seeking treatment have childhood and/or adult ADHD. Moreover, ADHD was overrepresented in adults with CUD compared to other substance use disorder patients seeking treatment. The importance in treating CUD individuals who also have ADHD is underscored by findings demonstrating that individuals with co-occurring ADHD and substance use disorders are a particularly intractable group: they exhibit earlier onset of use, more severe use, a more complicated pattern of remission/relapse, and poorer treatment outcomes relative to those without ADHD. Yet, to date, ADHD individuals with CUD have not been adequately studied. We have found that in our treatment research studies targeting cannabis dependence that a substantial percentage (35%) have screened positive for adult ADHD, rates that are higher than participants in our cocaine use disorder clinical trial and almost 8x greater than rates found in the general population (Kessler et al., 2006; Volkow et al., 2014). Thus, this appears to be a sizable cannabis-abusing group warranting much greater clinical attention than they are currently receiving.

While numerous studies have found that greater impulsivity is associated with poorer treatment outcome, particularly among those with ADHD, we will explore whether reduction in impulsivity is associated with less marijuana use. Further, we will assess sleep quality, a factor that might degrade the positive effects of medication treatment. While the administration of stimulants to active substance abusers remains controversial, a growing literature demonstrate that they can be given safely and at higher doses are effective in treating ADHD and stimulant use disorders. We would contend that if this study produces promising results, it will help be innovative in that it will inform clinical practice among a significant subgroup of patients seeking treatment for their CUD.

This proposal would be, to our knowledge, the first pharmacologic trial targeting individuals with CUD who also have ADHD, a group that represents approximately one-third of CUD individuals seeking treatment. The goal is to demonstrate feasibility, tolerability, and estimate effect size for purposes of planning future more definitive trials. Because of our team's extensive experience in working with stimulant medication in treating ADHD in cocaine-dependent populations, the large effect size of amphetamine in treating adult ADHD, and notable reduction in cocaine use and ADHD symptoms in cocaine-dependent ADHD adults, we will explore the efficacy of Adderall-XR (MAS-XR) for the treatment of cannabis use disorder and ADHD.

### **Specific Aims and Hypotheses**

Specific Aims and Hypotheses

**Primary Aim**: To determine among CUD individuals with ADHD whether MAS-XR is superior to placebo in: 1) promoting abstinence from cannabis use, and 2) reducing ADHD symptoms by at least 30% at the end of the maintenance phase.

- **Primary Hypothesis**: MAS-XR will be superior to placebo in promoting consecutive abstinence from marijuana use in the last 2 weeks of the study.
- **Hypothesis 2**: MAS-XR will be superior to placebo in promoting a 30% decrease of ADHD symptoms at the end of the study. The effect of treatment on both primary outcomes will be examined using logistic regressions adjusted for appropriate covariates which are known to be associated with each of the primary outcomes, respectively.

# Protocol Summary Form 7280 Levin, Frances

## NEWYORK STATE PSYCHIATRIC INSTITUTE INSTITUTIONAL REVIEW BOARD

**Secondary Aim**: To determine if MAS-XR is superior to placebo in secondary outcomes across key domains including: 1) other cannabis use outcomes; 2) other ADHD outcome measures; 3) neuropsychological traits associated with ADHD and substance use disorder, including measures of attention, memory, and impulsivity; 4) psychosocial functioning and mood outcomes; and 5) tolerability and retention.

- **Hypothesis 3**: Treatment will be superior to placebo in: a) reducing quantity of marijuana use, b) reducing the mean number of using days per week, and c) reducing symptoms of THC withdrawal.
- **Hypothesis 4**: Treatment will be superior to placebo in: a) reducing the percentage of individuals with CGI≤ 2, b) reducing the mean change from baseline in CAARS and AISRS
- **Hypothesis 5**: Treatment will be superior to placebo in reducing deficits in neuropsychological measures of impulsivity and attention
- **Hypothesis 6**: Treatment will be superior to placebo in: a) improving psychosocial functioning and quality of life, and b) reducing mood scores
- Hypothesis 7: Treatment will be superior to placebo in: a) participant retention and b) increasing time to drop-out. Patients in treatment will achieve a c) maximum tolerated dose of 80 mg on average, and d) will only demonstrate mild to moderate side effects. The secondary hypothesizes will be analyzed using generalized mixed effect models with appropriate link function (identity for continuous outcomes, binary for dichotomous outcomes), where participant will be treated as a random factor. Longitudinal outcomes will be analyzed similarly with generalized mixed effect models with time as fixed effect and GEE structure to model the within participant over-time correlations as autoregressive AR(1) process. Time to dropout will be analyzed using survival analyses and Kaplan-Meier method.

To test the hypothesis related to tolerability outcome, an average maximum tolerated dose achieved across all participants will be computed with appropriate 95% confidence interval. If the confidence interval includes 80 mg, we can conclude that the average overall achieved maximum dose is not significantly different than desired 80 mg. Similar analyses will be carried out for side effect outcomes.

**Exploratory Aim**: We will explore whether the reduction in ADHD symptoms (e.g. impulsivity, inattention) and sleep quality mediates the effect of treatment on cannabis use.

• Exploratory mediation hypothesis: Reduction in ADHD symptoms, change in impulsivity, change in sleep quality and other cognitive deficits will be tested as mediators of the relationship between treatment and cannabis use using the Baron and Kenny mediation framework.

### **Description of Subject Population**

#### Sample #1

Specify subject population

Protocol Summary Form 7280 Levin, Frances

Adults with CUD and ADHD

Number of completers required to accomplish study aims

25

Projected number of subjects who will be enrolled to obtain required number of completers

50

Age range of subject population

18-65

Gender, Racial and Ethnic Breakdown

We plan to randomization 40 participants into the study. Both males and females will be recruited. All eligible participants are accepted; however, past experience with recruitment for cannabis dependence suggests that the approximate gender distribution for this study will likely be 20% female and 80% male. Previous and ongoing marijuana studies at STARS have had samples comprised of approximately 50% Caucasians, and 50% ethnic minorities distributed as 24% African-American and 22% Hispanic-American, and 4% other. We anticipate a similar representation in this project. We will make every effort to recruit minority patients in order to ensure the generalizability of our findings to the overall treatment population. Description of subject population

We plan to enroll 50 participants into the study who meet criteria for current CUD and ADHD.

#### **Recruitment Procedures**

Describe settings where recruitment will occur

All screening and study procedures will occur at the Substance Treatment and Research Services (STARS) of the Division on Substance Abuse (STARS Downtown) situated on 3 Columbus Circle, 14th Floor, Suite 1403, NY, NY 10019.

How and by whom will subjects be approached and/or recruited?

Screening for this study will be covered by the Substance Treatment and Research Service (STARS) umbrella screening protocol #6582R (PI: John Mariani, MD). Trained research assistants and administrative assistants under the supervision of the principal investigator conduct the initial phone screening. Under protocol #6582R, patients who contact STARS interested in research trial participation are informed that they will be asked questions of a personal nature and asked to provide verbal consent for such questions. A "phone screen" form is completed by the phone screener, which asks basic demographic information, contact information (for scheduling purposes) and description of substance use to determine whether an inperson evaluation appointment is appropriate. Individuals are also informed that if they make an initial screening appointment this "phone screen" information will be forwarded to the clinician to facilitate the first meeting.

All patients will receive an explanation of the study risks, benefits, treatments, procedures, and option for alternative treatments. Patients who wish to participate will be asked to sign the treatment consent form following resolution of any questions and clear indication that they understand the nature of the study and consent form.

How will the study be advertised/publicized?

Levin, Frances

# NEW YORK STATE PSYCHIATRIC INSTITUTE INSTITUTIONAL REVIEW BOARD

We will recruit individuals with CUD and ADHD through newspapers, radio and public service announcements coordinated by the NYSPI Public Relations Office. This method has proven successful in several clinical trials at STARS. All advertisements will be sent to the Institutional Review Board for approval. The first phase of recruitment is a structured telephone interview when the initial contact is made. Individuals interested in receiving treatment for CUD and ADHD will be asked to come to STARS for additional screening as per protocol #6582R. Those patients who meet criteria for CUD and ADHD and all other inclusion/exclusion criteria will be asked if they are interested in participating in the study.

Do you have ads/recruitment material requiring review at this time?

No

Does this study involve a clinical trial?

Yes

YOU MUST REGISTER AT <u>ClinicalTrials.gov</u> IMMEDIATELY UPON RECEIPT OF IRB APPROVAL AND <u>PRIOR TO ENROLLMENT</u> OF THE FIRST SUBJECT. YOU WILL BE PROVIDED WITH A NCT REGISTRATION NUMBER ON REGISTRATION. PLEASE REVISE THIS SECTION OF THE PROTOCOL SUMMARY FORM TO INCLUDE THE NCT NUMBER AND RE-SUBMIT AS AN AMENDMENT TO THE IRB.

#### **Concurrent Research Studies**

Will subjects in this study participate in or be recruited from other studies?

Yes

Describe concurrent research involvement

Screening for this study will be covered by the Substance Treatment and Research Service (STARS) umbrella screening protocol #6582R (PI: John Mariani, MD). Trained research assistants and administrative assistants under the supervision of the principal investigator conduct the initial phone screening. Under protocol #6582R, patients who contact STARS interested in research trial participation are informed that they will be asked questions of a personal nature and asked to provide verbal consent for such questions. A "phone screen" form is completed by the phone screener, which asks basic demographic information, contact information (for scheduling purposes) and description of substance use to determine whether an inperson evaluation appointment is appropriate. Individuals are also informed that if they make an initial screening appointment this "phone screen" information will be forwarded to the clinician to facilitate the first meeting.

#### Inclusion/Exclusion Criteria

Name the subject group/sub sample
Adults with CUD and ADHD
Create or insert table to describe the inclusion criteria and methods to ascertain them

1) Individuals who meet criteria for cannabis use disorder (CUD) and report that marijuana is their primary drug of abuse report

2) Individuals must report using marijuana at least 5 days a week and have Participant

Levin, Frances

# NEWYORK STATE PSYCHIATRIC INSTITUTE INSTITUTIONAL REVIEW BOARD

a positive urine test for THC on the day of study entry self-report; urine drug screen Diagnostic Interview for 3) Individuals must meet DSM-5 criteria for adult ADHD ADHD in adults (DIVA) 4) Individuals who score > 22 on the AISRS scale **AISRS** Demographics 5) Individuals between the ages of 18-65 capable of giving informed ; MD consent and capable of complying with study procedures assessment 6) Women of child-bearing age will be included if they: a) are not pregnant, b) agree to use an effective method of contraception, c) agree not to become pregnant during the study and d) are not breastfeeding. To confirm this, urine pregnancy tests will be repeated every month after Self report; screening. Women will be provided a full explanation of the potential urine HCG dangers of pregnancy while taking MAS-XR. If a woman becomes pregnant, she will be taken off medication and continue standard treatment at STARS. At the end of the study, patients will be offered treatment at STARS until an appropriate referral can be made to a community clinic.

#### Create or insert table to describe the exclusion criteria and methods to ascertain them

| 1) Individuals meeting DSM-5 criteria for schizophrenia, schizoaffective illness, psychotic disorder other than transient psychosis due to drug abuse, current major depression, bipolar illness or psychiatric disorders (other than substance abuse) which require psychiatric intervention or would interfere with study participation | MINI;<br>psychiatric<br>evaluation |
|---|---|
| 2) Individuals who are medically unstable based on laboratory tests, electrocardiogram, medical history, physical examination that would make participation hazardous | Laborator<br>y tests;<br>medical<br>evaluation |
| 3) Use of synthetic cannabinoids in the past month and meeting CUD diagnosis based on synthetic cannabinoids use alone in the past year | MINI;<br>self report |
| 4) Individuals with liver enzyme function tests greater than 3 times normal | Laborator y tests |
| 5) Individuals with significant current suicidal risk | MINI;<br>psychiatric<br>evaluation |
| 6) Individuals with systolic blood pressure $>$ 140; diastolic blood pressure $>$ 90; pulse $>$ 100 | Vitals assessment |
| 7) Individuals who are cognitively impaired to impede study participation | Psychiatri c evaluation |
| 8) Nursing mothers and pregnant women | Self<br>report;<br>HCG |
| 9) Individuals who are physiologically dependent on any other drugs (excluding nicotine) that would require a medical intervention | MINI;<br>medical |

| | evaluation |
|---|---|
| 10) Individuals with known sensitivity/allergy to MAS-XR or amphetamir analogs | Self-<br>ne report;<br>medical<br>evaluation |
| 11) Individuals currently being prescribed psychotropic medication (include sleep medication) | Self- ling report; medical evaluation |
| 12) Individuals with history of seizures | Medical<br>history |
| 13) Individuals who are mandated to treatment | Self<br>report |
| 14) Individuals with a history of amphetamine <b>use disorders</b> , including amphetamines such as methamphetamine and MDMA. | MINI;<br>medical<br>evaluation |
| 15) Individuals with a current cocaine use disorder | al avaluation |

MINI; medical evaluation

#### Waiver of Consent/Authorization

Indicate if you are requesting any of the following consent waivers

Waiver of consent for use of records that include protected health information (a HIPAA waiver of Authorization)

No

Waiver or alteration of consent

No

Waiver of documentation of consent

No

Waiver of parental consent

No

#### **Consent Procedures**

Is eligibility screening for this study conducted under a different IRB protocol?

Yes

Indicate NYSPI IRB #

6582R

**Describe Study Consent Procedures** 

Screening for this study will be covered by the Substance Treatment and Research Service (STARS) umbrella screening protocol #6582R (PI: John Mariani, MD). Trained research assistants and administrative

NEWYORK STATE PSYCHIATRIC INSTITUTE
INSTITUTIONAL REVIEW BOARD

Levin, Frances

assistants under the supervision of the principal investigator conduct the initial phone screening. Under protocol #6582R, patients who contact STARS interested in research trial participation are informed that they will be asked questions of a personal nature and asked to provide verbal consent for such questions. A "phone screen" form is completed by the phone screener, which asks basic demographic information, contact information (for scheduling purposes) and description of substance use to determine whether an inperson evaluation appointment is appropriate. Individuals are also informed that if they make an initial screening appointment this "phone screen" information will be forwarded to the clinician to facilitate the first meeting.

Indicate which of the following are employed as a part of screening or main study consent procedures

✓ Consent Form

#### Persons designated to discuss and document consent

Select the names of persons designated to obtain consent/assent Brezing, Christina, MD
Dakwar, Elias, MD
Evans, Elizabeth, MD
Levin, Frances, MD
Luo, Sean, MD
Mariani, John, MD
Marino, Leslie, MD
Naqvi, Nasir, MD
Williams, Arthur
Type in the name(s) not found in the above list
Adam Bisaga, MD

### **Study Procedures**

Describe the procedures required for this study

#### General Design:

40 participants whom meet criteria for CUD and ADHD, and all other study inclusion and exclusion criteria (described above) will be randomized to the 12-week double-blind, placebo-controlled treatment trial. Patients will be randomized to receive either placebo or MAS-XR. Table 1 shows the overall design.

#### 1. Design Overview

The proposed protocol is a double-blind, placebo-controlled outpatient study of the safety and efficacy of Adderall-XR (MAS-XR) in the treatment of individuals with CUD and ADHD. We plan to randomize 40 patients in a 12-week trial. The primary objective of the study is to determine the efficacy of MAS-XR in promoting cannabis abstinence among individuals with CUD and in promoting a decrease of ADHD symptoms. The study will have a 1-week single-blind placebo lead-in phase; participants who are abstinent during this week, or noncompliant with study procedures, will not be randomized. After completion of the lead-in period (week 1), individuals will be randomized to MAS-XR or placebo, stratified by baseline

Protocol Summary Form 7280 Levin, Frances

ADHD rating, >35 or ≤35, at the end of week 1. Participants who are randomized to the medication arm will have their dose titrated to 80mg MAS-XR daily (over 2 weeks) and maintained on this dose for the subsequent 8 weeks. During week 12, participants will be tapered off of the medication (see Table 1. below). All participants will receive a supportive behavioral treatment that emphasizes study procedure adherence (Anton et al 2006; Johnson et al 2003b). Starting in week one, all patients will receive incentives for compliance with study procedures on an escalating reinforcement schedule similar to that developed previously (Budney et al 2000; 2006) and not contingent on urine results. The purpose of the lead-out is to blind patients to the exact point of medication discontinuation and to provide naturalistic data on the effects of medication discontinuation.

<u>Medication</u>: MAS-XR and matching placebo will be prepared by our pharmacy at the NYSPI packaged in matching gelatin capsules with lactose filler in each capsule. A PhD biostatistician at Columbia Univeristy, independent of the research team, will create the computer generated block design allociation sequence for the randomization. A non-blinded clinical psychologist at STARS allocates the randomization and informs the un-blinded NYSPI pharmacy who will then prepare the medications. At each weekly visit the psychiatrist orders the dose of double-blind medication for the coming week according to the schedule (shown in Table 2). The psychiatrist will adjust the dose according to tolerabillity. MAS-XR or matching placebo will be given in a fixed-flexible dose schedule with the MAS-XR dose titrated to 80mg per day or the maximum tolerated dose.

This dose was based on our experience with ADHD adults with cocaine use disorder. High placeboresponse rates can also obfuscate research findings. It has been our experience that even when patients have clear-cut diagnosis of ADHD, there is a subset of individuals who self-report ADHD improvement early on in treatment, prior to medication administration. Therefore, we will utilize the 1-week placebo lead-in period to stratify by baseline ADHD symptom severity, >35 or ≤35, prior to randomization and not randomize those who report no marijuana use during this lead-in period. In our prior cannabis trials we have used this procedure such that we did not randomize those who ceased using marijuana.

If a patient does experience any uncomfortable side effects, the dose will not be raised, and if necessary, the dose will be lowered. Patients will be encouraged to set a quit date three weeks after starting study medications (the end of the titration phase of MAS-XR). During week 12 patients on active medication will be tapered off MAS-XR.

We will evaluate the adequacy of the double-blind by asking patients which treatment drug they thing they are receiving. The blinded nurse will also be asked to report which drug s/he thinks each patient is taking. The research staff (i.e., therapist, nurse, research assistant and psychiatrist) that administers medications and/or conducts interviews and assessments will be blind to medication condition, urine toxicology results, and medication blood levels during the course of the 12-week trial. The non-blinded pharmacist and the non-blinded clinical psychologist will be the only ones who have access to this information during the trial. However, a sealed envelope will be kept in a locked office if the Principal Investigator needs to break the blind in an emergency situation. At the completion of the 12 week trial, or at the conclusion of the patient's involvement in the trial (if they do not complete all 12 weeks), patients will learn their treatment assignment.

Study medication will be over-capsulated with riboflavin to assess compliance using quantitative fluorometry. This non-harmful substance will allow the clinic to verify that the study medication is being taken correctly and absorbed by the body. The urine samples obtained twice a week will be examined for riboflavin. In addition, folic acid in the form of a 1 mg "pill" will be added to all placebo capsules in an attempt to improve the blind. The patient will receive up to 4 mg of folic acid daily. Patients will

Protocol Summary Form 7280 Levin, Frances

receive medication in non-childproof packaging. In the event that participants miss four consecutive days of medication, they will be given half the dose until their next scheduled study visit.

Medical Management Psychosocial Intervention: Phase II pharmacotherapy clinical trials should employ a psychosocial intervention to promote adherence to the study medication regimen and study visit schedule, without inflating the placebo response rate. The psychosocial intervention for this study will be Medical Management used for Project COMBINE (Anton et al., 2006), modified for cocaine dependence. All participants will have a manual-guided (Pettinati et al., 2005) supportive behavioral treatment session with the research psychiatrist each week. This psychosocial intervention facilitates compliance with study medication and other study procedures, promotes abstinence from marijuana and other substances, and encourages mutual-support group attendance. Dr. Mariani will provide ongoing supervision to other study physicians to prevent therapeutic drift. All study psychiatrists will be trained in providing Medical Management and refresher training sessions will be provided every 6 months. As director of Columbia's Substance Treatment and Research Service, Dr. Mariani has extensive experience conducting and supervising Medical Management and other similar medication adherence focused psychosocial intervention models.

<u>Patient Payments</u>: A voucher incentive system will be used to compensate patients for their time and travel and to encourage compliance with study procedures (visits and ratings). Patients will received \$10 for travel expenses at each visit (2x/week). Weekly return of medication bottles will receive \$10 each week.

Once entered into the study, patient can earn progressive weekly cash payments if they come to their study appointments, complete the required assessments, and provide a urine sample at each visit. Starting at \$2.50 for the first study visit, the value of the cash incentive for each subsequent consecutive visit is doubled to a maximum of \$25. Failure to attend study appointments, complete study assessments, and provide a urine sample will reset the value of cash incentives back to their initial \$2.50 from which the value can escalate again according to the same schedule. If an individuals attends all visits, they could earn \$563 in cash over a 12 week period. This reinforcement schedule occurs independently from the cash received for bottle return described above and cash compensation for travel.

<u>Assessment of Side Effects and Medication Compliance</u>: The research nurse and psychiatrist will query about side effects related to the study medication. Reported side effects and other treatment emergent events since the past visit will be recorded; additionally, the severity of the side effect/treatment emergent event, the action taken, and the continuation or resolution of the side effect/treatment emergent event will be documented.

a) Ongoing medical assessments. At each visit, the research nurse will monitor vital signs (heart rate and blood pressure) and inquire about medication-related side effects. Inability to tolerate medication side effects will result in the reduction or temporary discontinuation of study medications. Increases in blood pressure and heart rate considered unstable for two consecutive weeks (defined as SBP>140, DBP>90, sitting quietly HR>100) will result in the discontinuation of study medications. Unstable vital signs defined as SBP>160, DBP>110, sitting quietly HR>110 on any visit will result in immediate discontinuation from the study medications. The Side Effect Questionnaire consists of 2 parts: 1) self-reported side effects obtained by the nurse using an open format and 2) a checklist of symptoms rated from absent to severe, incorporating the major organ systems (e.g., gastrointestinal, neurological, cardiovascular). An ECG will be repeated at weeks 4 and 8 of the trial. An ECG and clinical blood work will also be repeated at the end of the study. Patients may be removed from the study if they repeatedly miss study visits.

Protocol Summary Form 7280 Levin, Frances

The research psychiatrist will meet with the patient once a week. At each weekly visit, s/he will discuss side effects of medication, review the Side Effect Questionnaire, will evaluate all reported vital signs and review cardiac risks to determine whether the dose is being tolerated, and assess substance use trends for clinical worsening. Cardiac risks will be documented in a structured progress note. If blood pressure and heart rate are consistently above cut-off levels as described above then the medication dose will be lowered or discontinued. If clinically indicated (e.g., side effects are not tolerable, chest pains, fainting, arrhythmias), the research psychiatrist will discontinue the medication. All participants will be re-consented between weeks 5-7 regarding anticipated risks and benefits to continued medication treatment. Participant response will be documented in the participant's record/chart.

b) <u>Urine Riboflavin</u>: A patients' compliance with respect to study medication will be monitored in two ways, by presence of riboflavin and pill count. The presence of riboflavin in a patients urine samples will be checked twice per week; the urine samples will be examined for riboflavin which will signifying the consumption of the study capsules. The absence of riboflavin in a patient's urine will not result in termination of a patient's involvement in the study. Secondly, medication compliance will be monitored by pill count on the medication bottles returned by the patient.

You can upload charts or diagrams if any table 1 study design.pdf medication titration schedule-table 2.pdf

### **Criteria for Early Discontinuation**

Criteria for Early Discontinuation

#### **Study Discontinuation**

Participants whose substance abuse significantly worsens during the course of treatment will be removed and treated clinically. If necessary, a referral for inpatient treatment will be made. This involves clinical judgment on the part of the treating psychiatrist(s) who are experienced with this population. This does not include transient modest worsening of drug use since substance dependence is a chronic relapsing condition. If more intensive treatment is deemed necessary, the participant will be offered continued weekly meetings with the physician until an appropriate referral can be made.

Drop-out criteria during the screening and study period include:

- 1) participant developing serious psychiatric symptoms (ADHD) as indicated by a Clinical Global Impression (CGI) improvement score of 6 (much worse than baseline) or greater for 2 consecutive weeks 2) participant's continued cannabis **use disorder**, even if improved from baseline, places him/her at risk for self-destructive behavior or other harm as indicated by a CGI improvement score of 6 (much worse than baseline) or greater for 2 consecutive weeks
- 3) female participant becoming pregnant as assessed by monthly urine pregnancy testing will result in cessation of the medication component but the option of continued participation in the trial and behavior therapy component.

Acute THC dosing can produce rises in blood pressure and heart rate, whereas chronic use may produce cardiovascular tolerance and rebound elevations in blood pressure/heart rate during cannabis withdrawal.

Protocol Summary Form 7280 Levin, Frances

Addition of amphetamine may increase these elevations further. Further, while we exclude individuals who have any history of a psychotic disorder or bipolar illness, it is possible that amphetamines, in addition to ongoing cannabis use, might elicit psychosis among individuals with underlying vulnerability. To address these safety concerns we will closely monitor patients throughout the trial for any evidence of cardiovascular problems or emerging psychosis and address this accordingly, as outlined in the DSMP. If we have any cardiovascular concerns based on our close weekly monitoring, we will consult with our cardiologist, Dr. Angelo Biviano. We have worked with him for close to a decade and he is well-acquainted with our outpatient clinical trials that test stimulant medications. Study medication discontinuation during the screening and study period will occur in the following instances:

- 1) If the patient develops signs of cardiovascular instability: weekly vital signs and clinical evaluation; pulse at rest > 100 or Blood Pressure at rest > 140/90 mm Hg for more than 2 weeks or SBP>160, DBP>110, HR>110 sitting quietly after being at the clinic for a period of time will result in immediate discontinuation of study medications
- 2) Cardiac risks as defined as cardiovascular chest pain, fainting or arrhythmias.

If a participant needs to be discontinued from study participation, he or she will be given the opportunity to continue with therapy as provided in the study, and treated clinically by the study psychiatrist or referred to a more appropriate level of care as needed.

#### **Blood and other Biological Samples**

Please create or insert a table describing the proposed collection of blood or other biological specimens

Approximately 20 ml of blood (4 teaspoons) will be drawn at the time of baseline assessment and study completion for routine analyses (hematology, blood chemistry (including liver function tests, chem-7, glucose, complete blood count), urinalysis, and blood pregnancy test for women). They may be repeated during the study if clinically indicated. Approximately, 40 ml of blood will be drawn overall (i.e., baseline and study completion =  $2 \times 20 \text{ ml} = 40 \text{ ml}$ ).

Quantitative urine toxicology screens for THC with Creatinine will be conducted at each visit (2 per week) and serve as an objective marker of current cannabis use. Quantitative toxicology for amphetamine and methylphenidate will be conducted every visit beginning in week 2.

HIV testing will be offered in order to determine the HIV status of all possible participants; participants may refuse if they do not want to be tested. Nursing staff will provide Pre and Post-test counselling to assist participants with any HIV+ results. Pre-HIV test counselling discusses the possibilities of a HIV+ test and the procedures after a positive HIV test is found. Post-HIV counselling assesses for suicidal and/or homicidal ideation, along with domestic violence issues. If a person tests positive for HIV, the research psychiatrist on staff with be notified and will do a secondary evaluation for necessity of immediate psychiatric care. Additionally the nursing staff will notify the department of health and provide a list of referrals for follow-up care.

A confirmatory HIV test will not routinely be done due to the accuracy of the saliva quick test, however if a participant tests positive using the saliva quick test a confirmatory blood test will immediately be done.

#### **Assessment Instruments**

Create a table or give a brief description of the instruments that will be used for assessment Screening: Psychiatric and substance use information will be obtained in the structured screening interview. The following evaluations will be used to determine whether a patient is appropriate for study participation. These data will be collected during the initial interviews and will cover inclusion/exclusion criteria. Additionally, a brief description of the study will be provided to eligible subjects to determine if the subject is interested in participating. If so, then informed consent will be obtained. Full screening will be completed within 1-2 weeks. The majority of measures in this treatment study are standard measures. Treatment Study Screening Procedures:

<u>Initial contact and interview</u>: The initial contact will include a brief interview to cover inclusion/exclusion criteria and a brief description of the study will be given to the patient to determine if the patient is interested in participating. If the patient is interested then an informed screening consent will be signed by the patient and witnessed by a member of the research staff.

Medical aspects: Patients will receive a full physical examination and an ECG before admission. Laboratory tests will include: hematology, blood chemistry (including liver function tests, chem-7, glucose, complete blood count, urinalysis, and blood pregnancy test for women)(45 minutes). An ECG will be repeated at weeks 4 and 8 of the trial. Patients will receive another physical examination and an ECG at end of study. Urine will be collected and tested for substances of abuse, twice weekly for the duration of the study. Demographic information: Patients will complete a Demographic Form, Medical and Psychiatric History Form, and Family Medical and Psychiatric History Form. These self-report forms provide data on age, race, socioeconomic status, marital status, educational and occupational levels, significant medical history, and current/history of major psychiatric disorder in the patient and his/her first-degree relatives. Patients will also complete a Locator Form so that they can be contacted for follow-up (30 minutes).

Please attach copies, unless standard instruments are used study assessments 4-11-16.pdf

### Off label and investigational use of drugs/devices

Choose from the following that will be applicable to your study

Urug

Select the number of drugs used in this study

#### Drug #1

Name of the drug Extended-release mixed amphetamine salt

# Protocol Summary Form 7280 Levin, Frances

### NEW YORK STATE PSYCHIATRIC INSTITUTE INSTITUTIONAL REVIEW BOARD

Manufacturer and other information

Other name: Adderall-XR® Manufacturer: Shire and Teva

Approval Status
IND is approved
IND#
79322
Who holds the IND/IND sponsor?
IND is held by PI/CU Investigator
Levin, Frances, MD

### **Research Related Delay to Treatment**

Will research procedures result in a delay to treatment?
Yes
Maximum duration of delay to any treatment
Once screening is completed, there is no delay for study entry for eligible patients.

The patient should receive treatment medication within 2-3 weeks after the initial screening evaluation if they have been randomized to the active medication arm. Those assigned to the placebo group will not receive active medication, but will receive medical management therapy within 2 weeks after the initial screening evaluation. Medical management therapy is an abstinence-focused supportive psychotherapy condition developed for substance use disorder pharmacotherapy clinical trials. Medical management therapy approximates the level of support of abstinence that patients would expect to receive in community treatment (general support of abstinence, tying improvement to reduction or cessation of drug use, referral to 12-step programs, etc.)

Maximum duration of delay to standard care or treatment of known efficacy
Because the screening procedure sometimes requires 2-3 meetings, individuals may not begin medical management therapy until 2-3 weeks after their initial screening evaluation for the study. Medical management therapy will start during the single-blind lead-in phase.

Treatment to be provided at the end of the study

At the conclusion of the 12-week protocol, the participants will be offered supportive therapy for at least one additional month or until an appropriate referral for on-going treatment is made.

If a patient was on active medications and they were shown to be beneficial, they will be given an appropriate referral for ongoing treatment.

#### **Clinical Treatment Alternatives**

Protocol Summary Form 7280 Levin, Frances

#### Clinical treatment alternatives

Individuals do not have to participate in this study to receive treatment for their cannabis use disorder and ADHD. Stimulant medication therapies, such as methylphenidate (Ritalin) as well as certain psychotherapy methods, may be helpful in treating the symptoms of ADHD. Although there are no accepted pharmacotherapies for the treatment of CUD. Psychotherapeutic approaches are commonly used for encouraging reduction in use or abstinence of drugs of abuse in general. These approaches include motivational enhancement, cognitive-behavioral therapy, 12-step facilitation, and other methods. Alternatives treatment settings for substance abuse include drug free outpatient treatment, inpatient detoxification, or residential treatment. Patients are informed that they may request referral for other treatment options. In addition, participants may withdraw from this study at any time and request referrals for other treatment options.

#### Risks/Discomforts/Inconveniences

Risks that could be encountered during the study period

#### **Potential Risks**

There are several sources and types of risk. Physical risks are those associated with obtaining blood samples (which may leave bruises) and medication administration. Psychological and social risks include revelation of sensitive material. Legal risks, not associated with the study per se, are inherent in the behavior of illicit drug use. The primary source of study related risks in clinical trials of medications stem from the medication itself. The following summarizes relevant information from the FDA approved prescribing information for MAS-XR.

MAS-XR: Amphetamine analog effects, benefits, and risks are extremely well understood. We recently completed a study using MAS-XR for adults with cocaine use disorder and ADHD. In addition, there is an extensive literature using amphetamines for the treatment of child and adult ADHD. Moreover, there is a worldwide replacement literature for amphetamine dependence; the cumulative data indicate comparatively low risk and the potential for considerable benefit. Still, risks are clear and can occur singly as the result of the medication itself, from interactions, or from additive effects in patients who abuse marijuana while receiving a therapeutic regimen.

Risks of oral amphetamines include nervousness, insomnia, blood pressure increases or decreases, gastrointestinal distress, weight loss and several forms of dermatitis. Side effects can be reduced or eliminated by lowering or discontinuing the medication. More severe effects include possible cardiovascular toxicity, particularly arrhythmias, excessive blood pressure elevation and the behavioral consequences of excessive CNS stimulation particularly sleep disturbance. Paranoid delusions, hallucinations, aggressive behavior, panic, anxiety, and a period of post drug depression are possible. Stroke and convulsions, although possible, are extremely unlikely at the doses used and in the population studied. Serious risk will be minimized by careful screening and dosing. No severe adverse events have been noted in previous studies and the medication appears to be well tolerated. The risk of abuse is of concern with the administration of amphetamine but is substantially lowered by administering extended release preparations. Although amphetamines have been prescribed for over 4 decades and no clear teratogenic risks have been described, it cannot be assumed that it is safe to administer during pregnancy. Female participants will be required to use adequate methods of birth control (condom with spermicide, diaphragm with spermicide, birth control pills). Serum pregnancy tests will be evaluated at baseline and monthly throughout the trial.

Participants may be at greater risk if they self-administer other drugs that interact with the study

Protocol Summary Form 7280 Levin, Frances

medications. Participants in these studies are identified users of marijuana and possibly other drugs. To the extent that they do not reduce or eliminate other drug use, risk may increase. Some of these risks are known others are of uncertain magnitude. In prior and ongoing studies that we are conducting with amphetamine analogs, no serious problems have emerged.

Female participants will be required to use adequate methods of birth control (condom with spermicide, diaphragm with spermicide, birth control pills). Urine pregnancy tests will be evaluated at baseline and monthly throughout the trial.

Finally, potential legal risks for these participants who use illegal drugs are addressed. Participants are advised to keep private materials related to the study. A certificate of confidentiality will be obtained.

As one progresses through the treatment study, depressive symptoms may emerge as a result of participants using marijuana or being unable to stop using. Depressive symptoms will be monitored once a month using the Hamilton Depression Scale.

The structured interviews, rating scales, and questionnaires should add no physical risk. The major disadvantage is the time required to complete them and that some of the questions might be embarrassing to patients. Our past experience with these measures indicates that they are acceptable to participants. However, some people have found them uncomfortable and/or tiring because the interviews/assessments are long and of a personal nature. Patients are informed that they may refuse to answer any questions and may ask to stop at any time. If participants become upset during the interviews/assessments, assistance will be made available to them.

Risks of Diversion The risks of stimulant diversion are small but not negligent. The SAMHSA National Survey on Drug Use and Health collects data on a broad array of substances of abuse, including non-medical use of prescription stimulants. For 2010, nonmedical stimulant use was 0.4%. While not insignificant, it is substantially lower than nonmedical use of tranquilizers or pain medication. The risk of abuse is of concern with the administration of amphetamine but is substantially lowered by administering extended release preparations. Nevertheless we will take several precautions to minimize the risks of abuse and/or diversion of MAS-XR. MAS-XR will be provided on a weekly basis and will contain riboflavin. Patients who are found to abuse/divert their study medication will be taken off their study medication. Describe procedures for minimizing risks

#### **Procedures for Risk Minimization**

The exclusion criteria are designed to minimize the medical and psychiatric risks to participants as discussed above, including risks of adverse events and side effects such as intoxication. Pregnant or lactating women or those not practicing reliable birth control methods are excluded. Patients are instructed to inform their psychiatrist immediately if they suspect they may be pregnant, and urine HCG is monitored monthly during the trial.

Patients with histories of psychotic illness other than transient drug-related psychosis that in the investigator's judgment are unstable or would be disrupted by study medication will be excluded. During the study, Dr. Levin, along with the clinic staff will coordinate clinical care. Additionally, the treating psychiatrist monitors participants' mental status weekly.

The baseline medical evaluation includes physical examination, blood chemistry profile (including liver function tests, chem-7, glucose, complete blood count, urinalysis, HCG) and electrocardiogram (ECG) is designed along with clinical history to detect chronic and unstable medical illnesses.

History of allergic or adverse reactions to MAS-XR is exclusionary. Participants with significant suicide risk at the time of initial evaluation or history of serious suicide attempt will be excluded and referred for

Protocol Summary Form 7280 Levin, Frances

appropriate non-research treatment. Participants will be examined for suicidal ideation and risk during their weekly visits with the research psychiatrist and participants who develop a significant risk during the trial will be removed from the study and treated as clinically indicated.

In order to minimize the risk associated with the study medication, vital signs (heart rate and blood pressure) and medication-related side effects will be monitored by the research nurse (or psychiatrist) twice a week. At each weekly visit the psychiatrist will discuss side effects of medication, review the Side Effect Questionnaire, will evaluate all reported vital signs and review cardiac risks to determine whether the dose is being tolerated. Inability to tolerate medication side effects will result in the reduction or temporary discontinuation of study medications. Further, we will have participants come for a post-taper study visit approximately 7-10 days after the last dose of MAS-XR to ensure that they are not experiencing any untoward effects and collect final study measures. If we cannot get them to attend the clinic we will attempt to garner information over the phone.

A calibrated fluorometer will be used to test for riboflavin in the urine. For many years our group has been adding riboflavin to our medication capsules to assess for medication adherence. However, our group found that the visual determination of the presence/absence of riboflavin using UV lights was woefully inaccurate and could be improved by using a quantitative cut-off to determine the presence/absence of supplementary riboflavin (Herron et al. 2013). Thus we now have more accurate assessment for medication adherence.

#### Data and Safety Monitoring Plan

Patients are closely monitored throughout the trial as described above. Dr. Levin, the Principal Investigators on this study will be responsible for data and safety monitoring throughout the trial. In addition to weekly psychiatric visits, cardiovascular side effects and suicidal events will be monitored independently (i.e., no formal involvement with the study patients) by a Safety Monitoring Board consisting of Drs. Maria Oquendo, Evaristo Akerele, and Soteri Polydorou. They will review data provided by the Principal Investigators on an annual basis to assess the recruitment, progress, safety, adverse events, and serious adverse events associated with the study. Individuals on the Safety Monitoring Committee will be blind to the study medication but can be informed by the un-blinded pharmacist, if a study patient is on Medication "A" or Medication "B" with one group receiving active medication and the other group receiving placebo. In this way, they can observe any problematic trends associated with one of the "medications." If they deem necessary, they can also request to know whether or not the participant received active medication or placebo. If they believe that termination of the trial is warranted, the blind of all study patients will be broken. The SAEs and AEs will be reviewed by the DSMB on an annual and as-needed basis.

#### Patient Education

All patients will be informed of the possible side effects and risks enumerated above through extensive discussions with the research psychiatrist during the consent process. Patients will be warned that risks, as yet unknown, may occur when combining study medications with cocaine or with other street drugs or alcohol. Patients will give informed consent before entering the study and will be re-consented between weeks 5-7 regarding the anticipated risks and benefits of medication treatment. Patients are instructed to call us if any untoward effects occur and are given the phone number of our 24-hour answering service. One of the affiliated physicians is on call 24 hours per day to answer questions and handle clinical emergencies.

### **Methods to Protect Confidentiality**

Protocol Summary Form 7280 Levin, Frances

Describe methods to protect confidentiality

#### Confidentiality

A Certificate of Confidentiality will be acquired for this study from the National Institute on Drug Abuse to offer protection for the privacy of participants by protecting identifiable research information from forced disclosure (e.g., through a subpoena or court order). The Certificate of Confidentiality will allow investigators and others with access to research records to refuse to disclose information that could identify participants in any civil, criminal, administrative, legislative, or other proceeding, whether at the Federal, State, or local level. The Certificate of Confidentiality is granted for studies that collect information that, if disclosed, could damage participants' financial, employability, insurability, or reputation, or have other adverse consequences.

We use coded records (i.e. initials and numbers), store signed consent forms in a locked safe, and try, to the best of our ability to maintain confidentiality. Only coded records will be entered into the computer and the security of electronic data is ensured at the level of the server, the user, and the database. We do, however, point out to prospective patients, that we cannot assure that their drug histories and other personal records might not become known.

Will the study be conducted under a certificate of confidentiality?

Yes, we will apply for the Certificate of Confidentiality

#### **Direct Benefits to Subjects**

Direct Benefits to Subjects

Benefits to participants include a comprehensive medical and psychiatric assessment, and possible improvement in their symptoms of CUD and ADHD.

### **Compensation and/or Reimbursement**

Will compensation or reimbursement for expenses be offered to subjects?

Yes

Please describe and indicate total amount and schedule of payment(s).

Include justification for compensation amounts and indicate if there are bonus payments.

Study visits will occur twice a week. Patients will be reimbursed \$10 for transportation at each study visit (\$10/visit, with maximum of \$240 over 12 weeks). In some instances when patients take alternative transportation (i.e. driving to the clinic) they will be reimbursed up to \$20 in cash if they provide receipts for expenses such as tolls and parking. As described above, progressive cash incentives will be provided for study visit attendance and compliance with other study procedures. If a patient attended all visits during the 12 week study (which is highly unlikely), he/she could earn \$563. This reinforcement schedule occurs independently from the cash received for bottle return (which is an extra bonus that can total a maximum of \$120 over the 12 weeks) and compensation for travel (\$10/visit, with maximum of \$240 over 12 weeks).

### **Uploads**

Upload the entire grant application(s)
Upload copy(ies) of unbolded Consent Form(s)
CUD-ADHD cf unbolded 4-6-16.pdf
7280 IND-frl.pdf
Upload copy(ies) of bolded Consent Form(s)
Upload evidence of FDA IND approval(s)
Upload copy(ies) of the HIPAA form
PP2PDFPrepUEAuthorization 3-22-16.pdf
Upload any additional documents that may be related to this study
7280\_FB\_ProvApp\_04-13-16.pdf

#### References

#### References

- 1. Levin FR, Evans SM, Kleber HD. Prevalence of adult attention-deficit hyperactivity disorder among cocaine abusers seeking treatment. Drug and alcohol dependence. 1998;52(1):15-25. PubMed PMID: 9788002.
- 2. Schubiner H, Tzelepis A, Milberger S, Lockhart N, Kruger M, Kelley BJ, et al. Prevalence of attentiondeficit/hyperactivity disorder and conduct disorder among substance abusers. The Journal of clinical psychiatry. 2000;61(4):244-51. PubMed PMID: 10830144.
- 3. van Emmerik-van Oortmerssen K, van de Glind G, Koeter MW, Allsop S, Auriacombe M, Barta C, et al. Psychiatric comorbidity in treatment-seeking substance use disorder patients with and without attention deficit hyperactivity disorder: results of the IASP study. Addiction. 2014;109(2):262-72. doi:10.1111/add.12370. PubMed PMID: 24118292; PubMed Central PMCID: PMC4112562.
- 4. Kessler RC, Adler L, Barkley R, Biederman J, Conners CK, Demler O, et al. The prevalence and correlates of adult ADHD in the United States: results from the National Comorbidity Survey Replication. The American journal of psychiatry. 2006;163(4):716-23. PubMed PMID: 16585449.
- 5. van Emmerik-van Oortmerssen K, van de Glind G, van den Brink W, Smit F, Crunelle CL, Swets M, et al. Prevalence of attention-deficit hyperactivity disorder in substance use disorder patients: a metaanalysis and meta-regression analysis. Drug and alcohol dependence. 2012;122(1-2):11-9. PubMed PMID: 22209385.
- 6. Molina BS, Pelham WE, Jr. Attention-deficit/hyperactivity disorder and risk of substance use disorder: developmental considerations, potential pathways, and opportunities for research. Annual review of clinical psychology. 2014;10:607-39. Epub 2014/01/21. doi: 10.1146/annurev-clinpsy-032813-153722. PubMed PMID: 24437435; PubMed Central PMCID: PMCPmc4097844.
- 7. Koob GF. Neural mechanisms of drug reinforcement. Annals of the New York Academy of Sciences. 1992;654:171-91. PubMed PMID: 1632582.
- 8. Volkow ND, Wang GJ, Kollins SH, Wigal TL, Newcorn JH, Telang F, et al. Evaluating dopamine reward pathway in ADHD: clinical implications. Jama. 2009;302(10):1084-91. doi: 10.1001/jama.2009.1308. PubMed PMID: 19738093; PubMed Central PMCID: PMC2958516.
- 9. Ponce G, Hoenicka J, Rubio G, Ampuero I, Jimenez-Arriero MA, Rodriguez-Jimenez R, et al.

Levin, Frances

# NEW YORK STATE PSYCHIATRIC INSTITUTE INSTITUTIONAL REVIEW BOARD

Association between cannabinoid receptor gene (CNR1) and childhood attention deficit/hyperactivity disorder in Spanish male alcoholic patients. Molecular psychiatry. 2003;8(5):466-7. PubMed PMID: 12808424.

- 10. Arcos-Burgos M, Velez JI, Solomon BD, Muenke M. A common genetic network underlies substance use disorders and disruptive or externalizing disorders. Human genetics. 2012;131(6):917-29. Epub 2012/04/12. doi: 10.1007/s00439-012-1164-4. PubMed PMID: 22492058; PubMed Central PMCID: PMCPmc3351604.
- 11. Volkow ND, Fowler JS, Wang GJ, Swanson JM, Telang F. Dopamine in drug abuse and addiction: results of imaging studies and treatment implications. Arch Neurol. 2007;64(11):1575-9. PubMed PMID: 17998440.
- 12. Volkow ND, Wang GJ, Fowler JS, Tomasi D, Telang F, Baler R. Addiction: Decreased reward sensitivity and increased expectation sensitivity conspire to overwhelm the brain's control circuit. Bioessays. 2010;32(9):748-55. PubMed PMID: 20730946.
- 13. Dickstein SG, Bannon K, Castellanos FX, Milham MP. The neural correlates of attention deficit hyperactivity disorder: an ALE meta-analysis. Journal of child psychology and psychiatry, and allied disciplines. 2006;47(10):1051-62. PubMed PMID: 17073984.
- 14. Rubia K, Halari R, Smith AB, Mohammad M, Scott S, Brammer MJ. Shared and disorder-specific prefrontal abnormalities in boys with pure attention-deficit/hyperactivity disorder compared to boys with pure CD during interference inhibition and attention allocation. Journal of child psychology and psychiatry, and allied disciplines. 2009;50(6):669-78. PubMed PMID: 19236528.
- 15. Bickel WK. Discounting of delayed rewards as an endophenotype. Biological psychiatry. 2015;77(10):846-7. doi: 10.1016/j.biopsych.2015.03.003. PubMed PMID: 25925716.
- 16. Finn PR, Gunn RL, Gerst KR. The Effects of a Working Memory Load on Delay Discounting in Those with Externalizing Psychopathology. Clinical psychological science: a journal of the Association for Psychological Science. 2015;3(2):202-14. doi: 10.1177/2167702614542279. PubMed PMID: 25893146; PubMed Central PMCID: PMC4399809.
- 17. Urban NB, Slifstein M, Thompson JL, Xu X, Girgis RR, Raheja S, et al. Dopamine release in chronic cannabis users: a [11c]raclopride positron emission tomography study. Biological psychiatry. 2012;71(8):677-83. doi: 10.1016/j.biopsych.2011.12.018. PubMed PMID: 22290115; PubMed Central PMCID: PMC3314125.
- 18. Martinez D, Gil R, Slifstein M, Hwang DR, Huang Y, Perez A, et al. Alcohol dependence is associated with blunted dopamine transmission in the ventral striatum. Biological psychiatry. 2005;58(10):779-86. doi: 10.1016/j.biopsych.2005.04.044. PubMed PMID: 16018986.64
- 19. Ghazzaoui R, Abi-Dargham A. Imaging dopamine transmission parameters in cannabis dependence. Progress in neuro-psychopharmacology & biological psychiatry. 2014;52:28-32. doi: 10.1016/j.pnpbp.2013.10.013. PubMed PMID: 24513022.
- 20. Martinez D, Narendran R. Imaging neurotransmitter release by drugs of abuse. Current topics in behavioral neurosciences. 2010;3:219-45. doi: 10.1007/7854 2009 34. PubMed PMID: 21161755.
- 21. Volkow ND, Wang GJ, Telang F, Fowler JS, Alexoff D, Logan J, et al. Decreased dopamine brain reactivity in marijuana abusers is associated with negative emotionality and addiction severity. Proceedings of the National Academy of Sciences of the United States of America. 2014;111(30):E3149-56. doi: 10.1073/pnas.1411228111. PubMed PMID: 25024177; PubMed Central PMCID: PMC4121778.
- 22. Backman L, Nyberg L, Soveri A, Johansson J, Andersson M, Dahlin E, et al. Effects of working-memory training on striatal dopamine release. Science. 2011;333(6043):718. doi: 10.1126/science.1204978. PubMed PMID: 21817043.

Levin, Frances

### NEW YORK STATE PSYCHIATRIC INSTITUTE INSTITUTIONAL REVIEW BOARD

- 23. Sheffer CE, Christensen DR, Landes R, Carter LP, Jackson L, Bickel WK. Delay discounting rates: a strong prognostic indicator of smoking relapse. Addictive behaviors. 2014;39(11):1682-9. doi:
- 10.1016/j.addbeh.2014.04.019. PubMed PMID: 24878037; PubMed Central PMCID: PMC4316833.
- 24. Stanger C, Ryan SR, Fu H, Landes RD, Jones BA, Bickel WK, et al. Delay discounting predicts adolescent substance abuse treatment outcome. Experimental and clinical psychopharmacology. 2012;20(3):205-12. doi: 10.1037/a0026543. PubMed PMID: 22182419; PubMed Central PMCID: PMC3906638.
- 25. Carroll KM, Rounsaville BJ. History and significance of childhood attention deficit disorder in treatment seeking cocaine abusers. Compr Psychiatry. 1993;34(2):75-82. PubMed PMID: 8485984.
- 26. Levin FR, Evans SM, Vosburg SK, Horton T, Brooks D, Ng J. Impact of attention-deficit hyperactivity disorder and other psychopathology on treatment retention among cocaine abusers in a therapeutic community. Addictive behaviors. 2004;29(9):1875-82. PubMed PMID: 15530732.
- 27. Wise BK, Cuffe SP, Fischer T. Dual diagnosis and successful participation of adolescents in substance abuse treatment. Journal of substance abuse treatment. 2001;21(3):161-5. PubMed PMID: 11728790.
- 28. Stinson FS, Ruan WJ, Pickering R, Grant BF. Cannabis use disorders in the USA: prevalence, correlates and co-morbidity. Psychological medicine. 2006;36(10):1447-60. PubMed PMID: 16854249.
- 29. Simon V, Czobor P, Balint S, Meszaros A, Bitter I. Prevalence and correlates of adult attention-deficit hyperactivity disorder: meta-analysis. The British journal of psychiatry: the journal of mental science. 2009;194(3):204-11. PubMed PMID: 19252145.
- 30. Pettinati HM, Volpicelli JR, Kranzler HR, Luck G, Rukstalis MR, Cnaan A. Sertraline treatment for alcohol dependence: interactive effects of medication and alcoholic subtype. Alcoholism, clinical and experimental research. 2000;24(7):1041-9. PubMed PMID: 10924008.
- 31. Anderson AL, Reid MS, Li SH, Holmes T, Shemanski L, Slee A, et al. Modafinil for the treatment of cocaine dependence. Drug and alcohol dependence. 2009;104(1-2):133-9. PubMed PMID: 19560290.
- 32. Elkashef AM, Rawson RA, Anderson AL, Li SH, Holmes T, Smith EV, et al. Bupropion for the treatment of methamphetamine dependence. Neuropsychopharmacology: official publication of the American College of Neuropsychopharmacology. 2008;33(5):1162-70. PubMed PMID: 17581531.
- 33. Nunes EV, Levin FR. Treatment of depression in patients with alcohol or other drug dependence: a meta-analysis. Jama. 2004;291(15):1887-96. PubMed PMID: 15100209.
- 34. Cunill R, Castells X, Tobias A, Capella D. Pharmacological treatment of attention deficit hyperactivity disorder with co-morbid drug dependence. Journal of psychopharmacology. 2015;29(1):15-23. doi: 10.1177/0269881114544777. PubMed PMID: 25142405.
- 35. Levin FR, Mariani JJ. Co-Occurring addictive disorder and attention deficit/hyperactivity disorder. In: Ries RK, Fiellin DA, Miller SC, R. S, editors. Principles of Addiction Medicine: American Society of Addiction Medicine, 5th Edition. New York, NY: Lippincott Williams & Wilkins; 2014. p. 1365-84.
- 36. Nunes EV, Covey LS, Brigham G, Hu MC, Levin FR, Somoza EC, et al. Treating nicotine dependence by targeting attention-deficit/ hyperactivity disorder (ADHD) with OROS methylphenidate: the role of baseline ADHD severity and treatment response. The Journal of clinical psychiatry. 2013;74(10):983-90. doi: 10.4088/JCP.12m08155. PubMed PMID: 24229749; PubMed Central PMCID: PMC3946795.
- 37. Levin FR, Evans SM, Brooks DJ, Garawi F. Treatment of cocaine dependent treatment seekers with adult ADHD: double-blind comparison of methylphenidate and placebo. Drug and alcohol dependence. 2007;87(1):20-9. PubMed PMID: 16930863.
- 38. Tamm L, Epstein JN, Lisdahl KM, Molina B, Tapert S, Hinshaw SP, et al. Impact of ADHD and cannabis use on executive functioning in young adults. Drug and alcohol dependence. 2013;133(2):607-14. doi: 10.1016/j.drugalcdep.2013.08.001. PubMed PMID: 23992650; PubMed Central PMCID:

7280 Levin, Frances

### NEW YORK STATE PSYCHIATRIC INSTITUTE INSTITUTIONAL REVIEW BOARD

#### PMC3820098.

- 39. Konstenius M, Jayaram-Lindstrom N, Guterstam J, Beck O, Philips B, Franck J. Methylphenidate for attention deficit hyperactivity disorder and drug relapse in criminal offenders with substance dependence: a 24-week randomized placebo-controlled trial. Addiction. 2013. doi: 10.1111/add.12369. PubMed PMID: 24118269.65
- 40. Levin FR, Mariani JJ, Specker S, Mooney M, Mahony A, Brooks DJ, et al. Extended-Release Mixed Amphetamine Salts vs Placebo for Comorbid Adult Attention-Deficit/Hyperactivity Disorder and Cocaine Use Disorder: A Randomized Clinical Trial. JAMA psychiatry. 2015;72(6):593-602. doi:
- 10.1001/jamapsychiatry.2015.41. PubMed PMID: 25887096; PubMed Central PMCID: PMC4456227.
- 41. Faraone SV, Buitelaar J. Comparing the efficacy of stimulants for ADHD in children and adolescents using meta-analysis. Eur Child Adolesc Psychiatry. 2009;19(4):353-64. PubMed PMID: 19763664.
- 42. Calipari ES, Ferris MJ, Siciliano CA, Jones SR. Differential influence of dopamine transport rate on the potencies of cocaine, amphetamine, and methylphenidate. ACS chemical neuroscience. 2015;6(1):155-62. doi: 10.1021/cn500262x. PubMed PMID: 25474655.
- 43. Dyck LE, Boulton AA, Jones RS. A comparison of the effects of methylphenidate and amphetamine on the simultaneous release of radiolabelled dopamine and p- or m-tyramine from rat striatal slices. European journal of pharmacology. 1980;68(1):33-40. PubMed PMID: 7449832.
- 44. Clausen SB, Read SC, Tulloch SJ. Single- and multiple-dose pharmacokinetics of an oral mixed amphetamine salts extended-release formulation in adults. CNS spectrums. 2005;10(12 Suppl 20):6-15. PubMed PMID: 16344836.
- 45. Castaneda R, Levy R, Hardy M, Trujillo M. Long-acting stimulants for the treatment of attention-deficit disorder in cocaine-dependent adults. Psychiatric services. 2000;51(2):169-71. PubMed PMID:10654994.
- 46. Wilens TE, Gignac M, Swezey A, Monuteaux MC, Biederman J. Characteristics of adolescents and young adults with ADHD who divert or misuse their prescribed medications. Journal of the American Academy of Child and Adolescent Psychiatry. 2006;45(4):408-14. PubMed PMID: 16601645.
- 47. Weisler RH, Biederman J, Spencer TJ, Wilens TE, Faraone SV, Chrisman AK, et al. Mixed amphetamine salts extended-release in the treatment of adult ADHD: a randomized, controlled trial. CNS spectrums. 2006;11(8):625-39. PubMed PMID: 16871129.
- 48. Spencer T, Biederman J, Wilens T, Faraone S, Prince J, Gerard K, et al. Efficacy of a mixed amphetamine salts compound in adults with attention-deficit/hyperactivity disorder. Archives of general psychiatry. 2001;58(8):775-82. PubMed PMID: 11483144.
- 49. Levin FR, Mariani JJ, Specker S, Mooney M, Mahony A, Brooks DJ, et al. Mixed Amphetamine Salts-Extended Release (Adderall-XR®) for Adults with Attention-Deficit/Hyperactivity Disorder and Cocaine Dependence: A Randomized Double-blind, Placebo Controlled TrialAccepted.
- 50. Riggs PD, Winhusen T, Davies RD, Leimberger JD, Mikulich-Gilbertson S, Klein C, et al. Randomized controlled trial of osmotic-release methylphenidate with cognitive-behavioral therapy in adolescents with attention-deficit/hyperactivity disorder and substance use disorders. Journal of the American Academy of Child and Adolescent Psychiatry. 2011;50(9):903-14. doi: 10.1016/j.jaac.2011.06.010. PubMed PMID: 21871372; PubMed Central PMCID: PMC3164797.
- 51. Moeller FG, Dougherty DM, Barratt ES, Schmitz JM, Swann AC, Grabowski J. The impact of impulsivity on cocaine use and retention in treatment. Journal of substance abuse treatment. 2001;21(4):193-8. PubMed PMID: 11777668.
- 52. MacKillop J, Kahler CW. Delayed reward discounting predicts treatment response for heavy drinkers receiving smoking cessation treatment. Drug and alcohol dependence. 2009;104(3):197-203. doi: 10.1016/j.drugalcdep.2009.04.020. PubMed PMID: 19570621; PubMed Central PMCID: PMC2740648.

Levin, Frances

- 53. Levin FR, McDowell D, Evans SM, Nunes E, Akerele E, Donovan S, et al. Pharmacotherapy for marijuana dependence: a double-blind, placebo-controlled pilot study of divalproex sodium. The American journal on addictions / American Academy of Psychiatrists in Alcoholism and Addictions. 2004;13(1):21-32. PubMed PMID: 14766435.
- 54. Carpenter KM, McDowell D, Brooks DJ, Cheng WY, Levin FR. A preliminary trial: double-blind comparison of nefazodone, bupropion-SR, and placebo in the treatment of cannabis dependence. The American journal on addictions / American Academy of Psychiatrists in Alcoholism and Addictions. 2009;18(1):53-64. PubMed PMID: 19219666.
- 55. Levin FR, Mariani J, Brooks DJ, Pavlicova M, Nunes EV, Agosti V, et al. A randomized double-blind, placebo-controlled trial of venlafaxine-extended release for co-occurring cannabis dependence and depressive disorders. Addiction. 2013;108(6):1084-94. doi: 10.1111/add.12108. PubMed PMID: 23297841; PubMed Central PMCID: PMC3636166.
- 56. Levin FR, Mariani J, Brooks DJ, M. P, Cheng C, Nunes E. Dronabinol for the treatment of cannabis dependence: A randomized, double-blind, placebo-controlled trial. Drug and alcohol dependence. 2011;116(1-3):142-50.
- 57. Mariani J, Brooks D, Haney M, Levin FR. Quantification and Comparison of Marijuana Smoking Practices: Blunts, Joints, and Pipes. Drug and alcohol dependence. 2011.
- 58. van de Glind G, van den Brink W, Koeter MW, Carpentier PJ, van Emmerik-van Oortmerssen K, Kaye S, et al. Validity of the Adult ADHD Self-Report Scale (ASRS) as a screener for adult ADHD in treatment seeking substance use disorder patients. Drug and alcohol dependence. 2013;132(3):587-96. doi: 10.1016/j.drugalcdep.2013.04.010. PubMed PMID: 23660242.66
- 59. Dakwar E, Mahony A, Pavlicova M, Glass A, Brooks D, Mariani JJ, et al. The utility of attentiondeficit/hyperactivity disorder screening instruments in individuals seeking treatment for substance use disorders. The Journal of clinical psychiatry. 2012;73(11):e1372-8. doi: 10.4088/JCP.12m07895. PubMed PMID: 23218166; PubMed Central PMCID: PMC3627386.
- 60. Levin FR, Evans SM, McDowell DM, Brooks DJ, Nunes E. Bupropion treatment for cocaine abuse and adult attention-deficit/hyperactivity disorder. J Addict Dis. 2002;21(2):1-16. PubMed PMID: 11916368.
- 61. Levin FR, Evans SM, McDowell DM, Kleber HD. Methylphenidate treatment for cocaine abusers with adult attention-deficit/hyperactivity disorder: a pilot study. The Journal of clinical psychiatry. 1998;59(6):300-5. PubMed PMID: 9671342.
- 62. Notzon DP, Mariani J, Pavlicova MA, Glass A, Mahony A, Brooks DJ, et al. Mixed-amphetamine salts increase abstinence from marijuana in patients with co-occurring Attention-Deficit/Hyperactivity Disorder and cocaine dependence. Submitted.
- 63. Pettinati HM, Weiss RD, Dundon W, Miller WR, Donovan D, Ernst DB, et al. A structured approach to medical management: a psychosocial intervention to support pharmacotherapy in the treatment of alcohol dependence. J Stud Alcohol Suppl. 2005(15):170-8; discussion 68-9. PubMed PMID:16223068.
- 64. Winhusen TM, Somoza EC, Brigham GS, Liu DS, Green CA, Covey LS, et al. Impact of attentiondeficit/hyperactivity disorder (ADHD) treatment on smoking cessation intervention in ADHD smokers: a randomized, double-blind, placebo-controlled trial. The Journal of clinical psychiatry. 2010. PubMed PMID: 20492837.
- 65. Carroll KM, Kiluk BD, Nich C, DeVito EE, Decker S, LaPaglia D, et al. Toward empirical identification of a clinically meaningful indicator of treatment outcome: features of candidate indicators and evaluation of sensitivity to treatment effects and relationship to one year follow up cocaine use outcomes. Drug and alcohol dependence. 2014;137:3-19. doi: 10.1016/j.drugalcdep.2014.01.012. PubMed PMID:24556275; PubMed Central PMCID: PMC4042667.

#### Protocol Summary Form 7280 Levin, Frances

# NEW YORK STATE PSYCHIATRIC INSTITUTE INSTITUTIONAL REVIEW BOARD

- 66. Herron AJ, Mariani JJ, Pavlicova M, Parrinello CM, Bold KW, Levin FR, et al. Assessment of riboflavin as a tracer substance: comparison of a qualitative to a quantitative method of riboflavin measurement. Drug and alcohol dependence. 2013;128(1-2):77-82. doi: 10.1016/j.drugalcdep.2012.08.007. PubMed PMID: 22921475; PubMed Central PMCID: PMC3556739.
- 67. Solanto MV, Marks DJ, Wasserstein J, Mitchell K, Abikoff H, Alvir JM, et al. Efficacy of metacognitive therapy for adult ADHD. The American journal of psychiatry. 2010;167(8):958-68. PubMed PMID:20231319.
- 68. Levin FR, Evans SM, Brooks DJ, Kalbag AS, Garawi F, Nunes EV. Treatment of methadonemaintained patients with adult ADHD: double-blind comparison of methylphenidate, bupropion and placebo. Drug and alcohol dependence. 2006;81(2):137-48. PubMed PMID: 16102908.
- 69. MTPRG. Marijuana Treatment Project Research Group. Brief treatments for cannabis dependence: Findings from a randomized multisite trial. J Consult Clin Psychol. 2004;72:455-66.
- 70. Dennis M, Godley SH, Diamond G, Tims FM, Babor T, Donaldson J, et al. The Cannabis Youth Treatment (CYT) Study: main findings from two randomized trials. Journal of substance abuse treatment. 2004;27(3):197-213. PubMed PMID: 15501373.
- 71. Mariani JJ, Pavlicova M, Bisaga A, Nunes EV, Brooks DJ, Levin FR. Extended-release mixed amphetamine salts and topiramate for cocaine dependence: a randomized controlled trial. Biological psychiatry. 2012;72(11):950-6. doi: 10.1016/j.biopsych.2012.05.032. PubMed PMID: 22795453;PubMed Central PMCID: PMC3648884.
- 72. Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, et al. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. The Journal of clinical psychiatry. 1998;59 Suppl 20:22-33;quiz 4-57. PubMed PMID: 9881538.
- 73. Epstein JN, Johnson DE, Conners CK. Conner's Adult ADHD Diagnostic Interview for DSM-IV (CAADID). North Tonawanda, NY: Multi-Health Systems, Inc.; 2001.
- 74. Johnson BA, Ait-Daoud N, Roache JD. The COMBINE SAFTEE: a structured instrument for collecting adverse events adapted for clinical studies in the alcoholism field. J Stud Alcohol Suppl. 2005(15):157-67; discussion 40. Epub 2005/10/15. PubMed PMID: 16223067.
- 75. Litten R, Allen J. Measuring Alcohol Consumption: Psychosocial and Biochemical Methods. Totowa, NJ: The Humana Press Inc.; 1992. 41-72.
- 76. Budney AJ, Hughes JR, Moore BA, Novy PL. Marijuana abstinence effects in marijuana smokers maintained in their home environment. Archives of general psychiatry. 2001;58(10):917-24. PubMed PMID: 11576029.
- 77. Guy W. ECDEU Assessment Manual for Psychopharmacology. Rockville, MD: US Department of Health, Education, and Welfare; 1976.
- 78. Williams JB. A structured interview guide for the Hamilton Depression Rating Scale. Archives of general psychiatry. 1988;45(8):742-7. PubMed PMID: 3395203.
- 79. Buysse DJ, Reynolds CF, 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry research. 1989;28(2):193-213. PubMed PMID: 2748771.
- 80. Conners C, Erhardt JN, Sparrow E. Conner's Adult ADHD Rating Scale (CAARS). North Tonawanda, NY: Multi-Health Systems; 1999.
- 81. Spencer TJ, Adler LA, Meihua Q, Saylor KE, Brown TE, Holdnack JA, et al. Validation of the adult ADHD investigator symptom rating scale (AISRS). Journal of attention disorders. 2010;14(1):57-68.

doi:10.1177/1087054709347435. PubMed PMID: 19794135.

- 82. Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacology Bulletin. 1993;29(2):321-6.
- 83. Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995;51(6):768-74. PubMed PMID: 8778124.
- 84. Allen TJ, Moeller FG, Rhoades HM, Cherek DR. Impulsivity and history of drug dependence. Drug & Alcohol Dependence. 1998;50(2):137-45.
- 85. Coccaro EF, Kavoussi RJ, Sheline YI, Lish JD, Csernansky JG. Impulsive aggression in personality disorder correlates with tritiated paroxetine binding in the platelet. Archives of general psychiatry. 1996;53(6):531-6. PubMed PMID: 8639036.
- 86. Cherek DR, Moeller FG, Dougherty DM, Rhoades H. Studies of violent and nonviolent male parolees: II. Laboratory and psychometric measurements of impulsivity. Biological psychiatry. 1997;41(5):523-9. PubMed PMID: 9046984.
- 87. Dougherty DM, Moeller FG, Steinberg JL, Marsh DM, Hines SE, Bjork JM. Alcohol increases commission error rates for a continuous performance test. Alcoholism, clinical and experimental research. 1999;23(8):1342-51. PubMed PMID: 10470977.
- 88. Dougherty DM, Marsh DM, Mathias CW. Immediate and delayed memory tasks: a computerized behavioral measure of memory, attention, and impulsivity. Behav Res Methods Instrum Comput. 2002;34(3):391-8. PubMed PMID: 12395555.
- 89. Robles E, Vargas PA. Parameters of delay discounting assessment: number of trials, effort, and sequential effects. Behavioural processes. 2008;78(2):285-90. doi: 10.1016/j.beproc.2007.10.012. PubMed PMID: 18222614.
- 90. Wechsler D. Wechsler Adult Intelligence Scale® Third Edition (WAIS®-III). San Antonio, TX: Pearson; 1997.
- 91. Dougherty DM, Mathias CW, Marsh DM. GoStop Impulsivity Paradigm (Version 1.0) Manual. Neurobehavioral Research Laboratory and Clinical, University of Texas Health Science Center Houston, Texas, 2003.
- 92. Dubbert PM, King A, Rapp SR, Brief D, Martin JE, Lake M. Riboflavin as a tracer of medication compliance. J Behav Med. 1985;8(3):287-99. PubMed PMID: 4087291.
- 93. Rotnitzky A, Scharfstein D, Su TL, Robins JM. Methods for conducting sensitivity analysis of trials with potentially nonignorable competing causes of censoring. Biometrics. 2001;57:103-13.
- 94. Fuller R, Roth H, Long S. Compliance with disulfiram treatment of alcoholism. J Chronic Dis. 1983;36(2):161-70. PubMed PMID: 6337171.
- 95. Fuller RK, Branchey L, Brightwell DR, Derman RM, Emrick CD, Iber FL, et al. Disulfiram treatment of alcoholism. A Veterans Administration cooperative study. Jama. 1986;256(11):1449-55. PubMed PMID:3528541.
- 96. Del Boca FK, Kranzler HR, Brown J, Korner PF. Assessment of medication compliance in alcoholics through UV light detection of a riboflavin tracer. Alcoholism, clinical and experimental research. 1996;20(8):1412-7. PubMed PMID: 8947318.
- 97. Sobell LC, Sobell MB. Timeline follow-back: a technique for assessing self-reported alcohol consumption in Measuring Alcohol Consumption. Litten RZ, Allen AJ, editors. Totowa, New Jersey: Humana Press; 1992. 41-72 p.
- 98. Hawks RL, Chiang CN. Examples of specific drug assays. NIDA Res Monogr. 1986;73:84-112. PubMed PMID: 3127725.
- 99. Wigal SB. Efficacy and safety limitations of attention-deficit hyperactivity disorder pharmacotherapy in

Levin, Frances

NEW YORK STATE PSYCHIATRIC INSTITUTE
INSTITUTIONAL REVIEW BOARD

children and adults. CNS Drugs. 2009;23 Suppl 1:21-31. PubMed PMID: 19621975.

- 100. Grabowski J, Rhoades H, Stotts A, Cowan K, Kopecky C, Dougherty A, et al. Agonist-like or antagonistlike treatment for cocaine dependence with methadone for heroin dependence: two double-blind randomized clinical trials. Neuropsychopharmacology: official publication of the American College of Neuropsychopharmacology. 2004;29(5):969-81.
- 101. Herin DV, Grabowski J. Agonist treatment for stimulant abuse and dependence. In: Miller PM, Kavanagh D, editors. Translation of Addictions Sciences into Practice. New York, NY: Elsevier Science; 2007. p. 145-67.
- 102. Herin DV, Rush CR, Grabowski J. Agonist-like pharmacotherapy for stimulant dependence: Preclinical human laboratory, and clinical studies. Addict Reviews. 2010;2:76-100.
- 103. Benowitz NL, Jones RT. Cardiovascular effects of prolonged delta-9-tetrahydrocannabinol ingestion. Clinical pharmacology and therapeutics. 1975;18(3):287-97. PubMed PMID: 1164818. 68
- 104. Vandrey R, Umbricht A, Strain EC. Increased blood pressure after abrupt cessation of daily cannabis use. Journal of addiction medicine. 2011;5(1):16-20. PubMed PMID: 21359104.
- 105. Kessler RC, Lane M, Stang PE, Van Brunt DL. The prevalence and workplace costs of adult attention deficit hyperactivity disorder in a large manufacturing firm. Psychological medicine. 2009;39(1):137-47. PubMed PMID: 18423074.
- 106. Matza LS, Paramore C, Prasad M. A review of the economic burden of ADHD. Cost Eff Resour Alloc. 2005;3:5. PubMed PMID: 15946385.

Schedule of Study Assessments

| Measure | Screen<br>ing | Lead-<br>In | Double-Blind Trial Week | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | Post-<br>taper<br>visit |
| MINI DSM psychiatric assessment | X | | | | | | | | | | | | | |
| Study Termination Form | Report | | | | | On | | | | | | Occurrence | | |
| Marijuana Use Assessments | | | | | | | | | | | | | | |
| Time Line Follow SUD | X | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | x |
| Marijuana Withdrawal Checklist | x | XX | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | x |
| Quantitative Toxicology for THC with Creatinine | х | XX | xx | xx | xx | XX | xx | xx | xx | xx | xx | xx | xx | x |
| CGI-O for Substance Use | х | х | х | х | х | х | х | х | х | х | х | х | х | х |
| Sleep assessment | | | | | | | | | | | | | | х |
| Pittsburgh Sleep Quality Index | х | | | | Х | | | | х | | | | х | х |
| ADHD Assessments | | | | | | | | | | | | | | |
| DIVA (Diagnostic Interview for ADHD in Adults) | х | | | | | | | | | | | | | |
| AISRS | х | x | х | х | х | х | х | х | х | х | х | х | х | х |
| CAARS-Self | х | Х | | | х | | | | х | | | | х | х |
| CGI-O for ADHD Symptoms | х | х | х | х | Х | х | х | Х | х | х | Х | х | х | х |
| Cognitive Assessment | | | | | | | | | | | | | | |
| Barratt Impulsiveness | х | | | | | | | | | | | | | |
| Immediate and Delayed Memory | х | | | | | | х | | | | | | | |
| GoStop | х | | | | | | х | | | | | | | |
| Letter-Number Sequencing | х | | | | | | х | | | | | | | |
| Delay Discount Program | х | | | | | | х | | | | | | | |
| Other Psychiatric/Life | | | | | | | | | | | | | | |
| Assessments | | | | | | | | | | | | | | |
| Hamilton Depression. Scale | х | х | | | х | | | | х | | | | x | x |
| Quality of Life, Enjoyment, and | x | | | | | | x | | | | | | x | x |
| Satisfaction | | | | | | | | | | | | | | |
| Medical Assessment | | | | | | | | | | | | | | |
| Physical/Bloods | X | | | | | | | | | | | | х | |
| Nursing Assessment | х | XX | XX | XX | XX | xx | XX | XX | XX | XX | XX | XX | xx | |
| Serum HCG (Urine HCG except at | x | | | | x | | | | x | | | | x | |
| baseline) | | | | | | | | | | | | | | |
| Concomitant Meds Form | x | X | x | x | x | x | x | х | х | x | x | х | х | x |
| MDRU Adverse Event | | X | X | x | X | х | X | X | X | x | X | х | х | x |
| Serious Adverse Event | Report | | | | | on | | | | | | Occurrence | | x |
| Medication Compliance | | XX | xx | xx | xx | xx | xx | xx | XX | xx | xx | xx | xx | |
| 12 Lead ECG | X | | | | х | | | | Х | | | | X | |
| HIV Testing | х | | | | | | | | | | | | | |
| Adherence Assessment | | | | | | | | | | | | | | |
| Quantitative Toxicology for | | | XX | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx | |
| Amphetamine & | | | | | | | | | | | | | | |
| Methylphenidate | | | | | | | | | | | | | | |
| Bottle Return with pill count | х | X | X | X | X | х | X | х | X | X | х | х | х | |
| Riboflavin Fluorometry | X | X | X | X | X | X | X | X | X | X | X | X | X | |

Table 1. Overall study design

| | Week 1 | Weeks 2-3 | Weeks 4-11 | Week 12 |
|---|---|---|---|---|
| | Single-Blind<br>Placebo Lead-In | Induction Phase | Maintenance Phase | Taper Phase |
| Group 1 | Placebo | MAS-XR (2 weeks) | MAS-XR 80 mg daily | MAS-XR taper |
| Group 2 | Placebo | Placebo | Placebo | Placebo |

 Table 2. Medication Titration Schedule

| Placebo<br>Lead-In<br>(Week 1) | Randomization<br>(Day 1) | Week 2<br>Days 1-2 | Week<br>2<br>Days<br>3-4 | Week 2<br>Days<br>5-6 | Week 3<br>Days 7-<br>9 | Week3<br>Days 10-12 | Week 3<br>Day 13-14 | Weeks<br>4-11 | Week 12 |
|---|---|---|---|---|---|---|---|---|---|
| Lead-In<br>Phase | | | Maintenance Phase | Taper Phase | | | | | |
| Placebo<br>qAM | MAS-XR | MAS-XR<br>20<br>mg/day | MAS-XR 30<br>mg/day | MAS-XR<br>40<br>mg/day | MAS-XR<br>50<br>mg/day | MAS-XR<br>60 mg/day | MAS-XR<br>70 mg/day | MAS-XR<br>80 mg/day | MAS-XR<br>(taper) |
| Placebo<br>qAM | Placebo Group | Placebo<br>qAM. | Placebo<br>qAM | Placebo<br>qAM | Placebo<br>qAM | Placebo qAM | Placebo qAM | Placebo qAM | Placebo q AM |